CLINICAL TRIAL: NCT06258876
Title: Mise en Place et rétention en médecine générale d'un Programme de Prophylaxie pré-exposition du VIH
Brief Title: Human Immunodeficiency Virus Pre-exposure Prophylaxis Program in General Practice
Acronym: PrEPInTheCity
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220156
Record Dates: First submitted 2024-01-23; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Human Immunodeficiency Virus
Keywords: Pre-exposure Prophylaxis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an indication for PrEP: - Any patient presenting to a general medicine consultation for initial PrEP prescription or having previously received a hospital-initiated PrEP prescription, in a CEGGID (Centres gratuits d'information, de dépistage et de diagnostic), in a sexual health center, and not having had a PrEP prescription renewal for at least 4 months.
  OR
  - Any patient seen in a general medicine consultation with an indication for PrEP.
  Interventions: Other: PrEP in general practice

INTERVENTIONS:
Other: PrEP in general practice — Prescription and follow-up of PrEP in general practice

SUMMARY:
The Human Immunodeficiency Virus (HIV) epidemic persists in France, with approximately 6000 new cases per year. Various prevention tools against HIV exist, including condoms, regular testing, Post-Exposure Prophylaxis (PEP), HIV treatment for seropositive partners, single-use disposable injection equipment for drug use and pre-exposure prophylaxis (PrEP).

Continuous or on-demand PrEP with tenofovir disoproxil fumarate/emtricitabine has proven effective in reducing the risk of HIV infection. France was the first European country to authorize PrEP, leading to an unprecedented impact on seropositivity discovery rates in 2018, with a 7% decrease in new infections compared to 2017.

However, the effectiveness of PrEP can be hindered by challenges in retaining users within the healthcare system. According to the EPIPHARE report, which has been monitoring Truvada® or generic PrEP use since 2017, a substantial proportion of new users do not receive PrEP renewal in the first 6 months after initiation. Such early interruptions, increasing in frequency, affected around a quarter of individuals who initiated PrEP in the second half of 2021.

A recent study reported that these early interruptions have a significant detrimental impact on PrEP effectiveness in real life, especially among those under 30 years old and in socio-economic precarious situations.

The main barriers to PrEP adherence are multifactorial, including social precarity, limited PrEP access, and a low perception of HIV risk. To address this, in France, general practitioners have been authorized to issue initial PrEP prescriptions since June 1, 2021.

The future challenge is to increase PrEP use and optimize retention to combat the HIV epidemic, relying significantly on general medicine. The goal of our study is to broaden PrEP access by optimizing its initial prescription in general medicine and to assess user retention in PrEP care through the established partnership between general practitioners and patients.

The research will be conducted in collaboration between Saint Louis Hospital in the 10th arrondissement of Paris and general practitioners willing to participate in the study, located in the 3rd, 10th, 11th, 13th, and 19th arrondissements. Participating general practitioners may be in private practice, employed in health centers, or working in health houses.

As part of the study, general practitioners will receive training from the infectious diseases department of Saint-Louis and Lariboisière hospitals. This training will be both theoretical and practical, with the opportunity to attend initiation and follow-up PrEP consultations in the department. A dedicated phone line in the infectious diseases department of Saint Louis Hospital will be available for participating general practitioners seeking specialized advice. They will be encouraged to register as PrEP prescribers in their appointment scheduling software.

Patients will be informed of the study objectives and its process by the general practitioner, and their oral non-opposition will be collected.

Each inclusion consultation will last approximately 20-40 minutes, allowing the general practitioner to prescribe PrEP, conduct the usual care consultation, and collect clinical, demographic, socio-economic, lifestyle, medical history, and patient vaccination data on a dedicated data collection form.

The follow-up duration will be two years, with consultation frequency matching that of regular PrEP follow-ups, and data collection will occur at M6, M12, M18, and M24 using a dedicated data collection form.

Data collected during inclusion and follow-up consultations will be anonymized and integrated into the electronic Clinical Report Form. During each PrEP consultation (initiation and follow-up), general practitioners will provide patients with a PrEP prescription if the pre-PrEP biology report allows it (according to HAS (Haute Autorité de Santé) recommendations).

For patients who have not been attending consultations, a telephone survey will be offered to inquire about PrEP continuation and collect information on follow-up or reasons for stopping PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed and provided verbal non-opposition
* Patient not infected with HIV and confirmed negative for the detection of antibodies produced in response to the HIV virus within the last 7 days (Elisa test) or recognized as having a negative HIV viral load
* Patient presenting in a general medicine consultation for:

  1. Initial prescription of PrEP
  2. Renewal consultation for PrEP (previously provided in a hospital, CEGGID, or sexual health center) without a PrEP prescription renewal for at least 4 months
  3. Consultation for another reason in general medicine and the patient presents one or more indications for PrEP prophylaxis:

     1. Belonging to one of these risk groups :
* MSM (men who have sex with men)
* Transgender individuals having relationships with men
* Individuals from regions with a high HIV prevalence (sub-Saharan Africa, Caribbean, South America)
* Sex workers
* Injectable drug users
* Any individuals (men and women) whose sexual partners belong to these populations

  b) Individual situation of high HIV exposure:
* High number of partners
* Partner living with HIV with an uncontrolled or unknown viral load
* Non-use of condoms
* Exposure to sexual violence
* Documented history of sexually transmitted infections (STIs) (syphilis, Neisseria gonorrhea, Mycoplasma genitalium, Chlamydia trachomatis, acute hepatitis C) or use of post-exposure prophylaxis (PEP) in the last 12 months.
* Affiliated with a social security system (beneficiary or dependent).

Exclusion Criteria:

* Patient with a contraindication to PrEP:

  1. Renal insufficiency with creatinine clearance < 60 ml/min
  2. Hypersensitivity to the components of PrEP (tenofovir disoproxil, emtricitabine, or excipients of the product)
* Patient refusal to participate in the study
* Patient who received a renewal of the PrEP prescription less than 4 months ago
* Patient under guardianship, curatorship, or legal protection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any patient presenting to a general medicine consultation for initial PrEP prescription or having received a hospital-initiated PrEP prescription, in a CEGGID, in a sexual health center, and not having had a PrEP prescription renewal for at least 4 months. Also, any patient seen in a general medicine consultation with an indication for PrEP.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients still on PrEP | At 2 years
  Any patient having a general medicine consultation with a PrEP prescription between 21 and 27 months following the first PrEP prescription

SECONDARY OUTCOMES:
Percentage of Patients still on PrEP | At 6 months
  Defined as any patient who had a general medicine consultation with a PrEP prescription at 6 months following the first PrEP prescription.
Percentage of Patients still on PrEP | At 12 months
  Defined as any patient who had a general medicine consultation with a PrEP prescription at 12 months following the first PrEP prescription.
Percentage of Patients still on PrEP | At 18 months
  Defined as any patient who had a general medicine consultation with a PrEP prescription at 18 months following the first PrEP prescription.
Characteristics of PrEP-Using Populations Initiated in General Medicine | Up to 2 years
  It includes risk group, initiation modality (suggested by the general practitioner or at the patient's request)
Characteristics of HIV at-Risk Populations with Limited Access to PrEP | At baseline
  Assessing geographical origin, social protection, profession, social precarity (evaluated by EPICES (Evaluation of precariousness and health inequalities in health examination centers) score : 11 questions score. The score varies between 0 and 100, the higher the score, the more precarious the situation.
Characteristics of HIV at-Risk Populations with Limited Access to PrEP | At 2 years
  Assessing geographical origin, social protection, profession, social precarity (evaluated by EPICES (Evaluation of precariousness and health inequalities in health examination centers) score : 11 questions score. The score varies between 0 and 100, the higher the score, the more precarious the situation.
Factors Associated with PrEP Discontinuation | At 2 years
  Including PrEP-related toxicity, entering into a relationship, adherence difficulties, lack of social protection, geographical origin, profession, social precarity.
Factors Associated with Follow-Up Discontinuation | At 2 years
  Involving loss to follow-up, change of general practitioner, or change in prescription location.
Cumulative Incidence of Side Effects | At 2 years
  Assessing the overall occurrence of side effects over the study period.
Cumulative Incidence of HIV Infection Diagnoses | At 2 years
Cumulative Incidence of Sexually Transmitted Infection (STI) Diagnoses | At 2 years
Proportion of Patients for Whom PrEP Could Be Resumed After a Break of 4 Months or More | At 2 years
  Assessing the proportion of patients for whom PrEP was successfully resumed after a break of 4 months or longer.
Proportion of Participating Physicians in the Infectious Diseases Service Training | At 2 years
  Including a satisfaction survey for the training, and the number of monthly calls received by the hospital platform for prescription assistance.
Percentage of Patients still on PrEP among those who previously had a PrEP prescription | At 2 years
  Including those who received a hospital-initiated PrEP prescription, in a CEGGID, or in a sexual health center and had not had a PrEP prescription renewal for at least 4 months before inclusion in the study

IPD SHARING:
Plan to Share IPD: Undecided